CLINICAL TRIAL: NCT00173368
Title: Study of Endoscopic Sphincterotomy With Needle Knife Papillotome in Patients of Ampullary Impacted Stone
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700651
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-08

CONDITIONS: Choledocholithiasis; Endoscopy
Keywords: Sphincterotomy; needle knife; hemorrhage; complication
MeSH Terms: conditions — Choledocholithiasis; Hemorrhage

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Using a needle knife papillotome by an experienced endoscopist, endoscopic sphincterotomies were performed in difficult cannulation cases. In a prospectively collected database, we investigate the complications of those with ampullary impacted stone.

DETAILED DESCRIPTION:
The endoscopic sphincterotomy with needle knife papillotome is a well-established advanced endoscopic technique in difficult cannulation cases. Choledocholithiasis impacted at the ampulla of Vater is occasionally seen. Inflammed surrounding mucosa frequently accompanies. Whether sphincterotomy with a needle knife increases the bleeding complications is to be elucidated in this study.

ELIGIBILITY:
Inclusion Criteria:

* choledocholithiasis patients and an ampullary impacted stone

Exclusion Criteria:

* patients with liver cirrhosis , pregnancy, history of abdominal malignancy, bleeding diathesis, ileus, renal failure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-01; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Po Wang, MD, Study Chair — National Taiwan University Hospital